CLINICAL TRIAL: NCT03662269
Title: Indomethacin for Refractory Chronic Cough: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Indomethacin for Refractory Chronic Cough
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Kefang Lai, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YDMX02V2.0
Record Dates: First submitted 2018-08-31; First posted 2018-09-07 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Indomethacin; Omeprazole

STUDY DESIGN:
Intervention Model Description: a randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indomethacin treatment group (Experimental): indomethacin (75mg, bid) + omeprazole (20mg, qd)
  Interventions: Drug: indomethacin; Drug: Omeprazole
- placebo treatment group (Placebo Comparator): placebo (75mg, bid) + omeprazole (20mg, qd)
  Interventions: Drug: Placebo; Drug: Omeprazole

INTERVENTIONS:
Drug: indomethacin — indomethacin (75mg, bid, po, 14days)
  Other Names: Indometacin sustained-release capsules
  Arms: indomethacin treatment group
Drug: Placebo — placebo (75mg, bid, po, 14days)
  Arms: placebo treatment group
Drug: Omeprazole — placebo (20mg, qd, po, 14days)

SUMMARY:
Chronic cough is a common complain of patients in respiratory clinic and its global prevalence was up to 9.6%. Persistent cough of unexplained origin is a significant health issue that occurs in up to 5% to 10% of patients seeking medical assistance for a chronic cough and from 0% to 46% of patients referred to specialty cough clinics. Previous studies showed that sputum prostaglandin D2( PGD2) and prostaglandin E2 (PGE2) concentrations were significantly higher in chronic cough. And some research showed that Inhaled PGE2 /PGF2α /PGD2 / PGI2/ 6-oxo-PGF1a could induced cough. And PGE2 /PGF2α/PGI2/thromboxane A2 (TXA2) also increased the sensitivity of the cough reflex. All these five primary prostaglandins were synthesized though the metabolism of arachidonic acid via the cyclooxygenase pathway. Indomethacin is a strong inhibitor of cyclooxygenase , which decrease the level of prostaglandins in airway. The investigator's preliminary study showed that indomethacin could relieve cough and improve cough sensitivity of some patients with refractory cough. Therefore this randomized, double-blind, placebo-controlled trial were designed to investigate whether indomethacin can relive cough in patients with refractory cough and to explore the possible mechanism of indomethacin in improving cough in patients with refractory cough.

ELIGIBILITY:
Inclusion Criteria:

1）18 years old ≤ age ≤ 60 years old, male or female; 2）Chronic cough lasting more than 8 weeks as the sole or predominant symptom, without abnormalities on chest radiograph; 3）Chronic cough remains after investigation and supervised therapeutic trial(s) conducted according to "Clinical Practice Guidelines for Diagnosis and Management of Cough (2015)" 4）Cough VAS (0-100mm) ≥ 30 mm

Exclusion Criteria:

1. Patients had any contraindications to indomethacin;
2. Patients had active respiratory disease (such as chronic obstructive pulmonary Disease or untreated asthma), or moderate or above obstructive or restrictive or mixed pulmonary ventilation dysfunction;
3. Patients had a respiratory tract infection in the month before randomization;
4. Patients were taking an angiotensin-converting enzyme inhibitor;
5. Patient were pregnant or breastfeeding, or had impaired kidney function;
6. Current and recent smokers (<6 months' abstinence), or ex-smokers with more than 20 pack-years (20 cigarettes per pack).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Cough Severity | 1, 3, 7, 10, 14, 21day
  Outcome measure: Cough visual analogue scales (Cough VAS). Score range: 0-100mm (0 mean no cough, 100 represent that cough is the most severe in his/her life. Scoring higher on cough VAS mean more severe cough he/she has. )
Change of cough-specific-quality-of-life | 1, 14, 21 day
  Outcome measure: Leicester Cough Questionnaire (LCQ). Score range: 3-21 (Higher values represent a better outcome.)

SECONDARY OUTCOMES:
frequency of patients'coughs | 1, 7, 14 day
  Outcome measure: cough count in one hour
laryngeal dysfunction score | 1, 7, 14 day
  Outcome measure: Laryngeal dysfunction questionnaire (Higher score represent a better outcome)
cough reflex sensitivity | 1, 7, 14, 21 day
  Outcome measure: LogC5 of Capsaicin cough challenge

OTHER OUTCOMES:
change of airway arachidonic acid metabolism | 1, 7, 14, 21 day
  Concentration of PGE2, PGF2α, PGD2, 6-Keto-PGF1α, TXB2, leukotriene B4(LTB4) and cys-LTs in induced sputum

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol Statistical Analysis Plan (SAP)